CLINICAL TRIAL: NCT05658068
Title: Experimental Evaluation of a Multi-site Suicide Intervention for Youth During and After Residential Placement
Brief Title: Systems Aligning for Equity (SAFE) Spaces
Acronym: SAFE Spaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-FY2019-3228
Record Dates: First submitted 2022-12-01; First posted 2022-12-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Suicide; Mental Disorder; Mental Health; Burnout, Professional; Self Harm
MeSH Terms: conditions — Suicide; Mental Disorders; Psychological Well-Being; Burnout, Professional; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAFE Spaces training and coaching (Experimental): Staff in facilities assigned to this arm are offered the SAFE Spaces training and coaching model.
  Interventions: Behavioral: SAFE Spaces training and coaching
- Training as Usual (No Intervention): Staff in facilities assigned to this arm receive training as usual.

INTERVENTIONS:
Behavioral: SAFE Spaces training and coaching — Staff in facilities assigned to the intervention are eligible to receive evidence-based programming in suicide detection and prevention (Shield of Care; SOC) and wellness skill-building (Skills for Life) through training and personalized coaching. Multiple training sessions will be offered to small groups of staff in-person in residential facilities and paired with personalized in-person and virtual coaching.
  Arms: SAFE Spaces training and coaching

SUMMARY:
The goal of this 2-arm cluster randomized clinical trial is to test whether an evidence-based staff training and coaching model specifically designed as a response to legal system-involved youths' and frontline staff's mental health needs can improve the safety and suicide outcomes, mental health challenges, and wellness and facility climate for youth and staff in facilities assigned to the intervention condition. Staff in facilities assigned to the intervention are eligible to receive evidence-based programming in suicide detection and prevention (Shield of Care; SOC) and wellness skill-building (Skills for Life) through training and personalized coaching. Multiple training sessions will be offered to small groups of staff in-person in residential facilities and paired with personalized in-person and virtual coaching. Staff and youth in all facilities will be asked to complete periodic surveys assessing experiences in the facility, suicide and safety knowledge and risk, and their mental health and wellness. Researchers will compare outcomes of staff in youth in facilities assigned to the intervention compared to facilities in the training-as-usual condition.

ELIGIBILITY:
Inclusion Criteria:

* Placement in in ACS-run or contracted residential facilities enrolled in the study during the first 2 years of the intervention period
* Proficiency in English

Exclusion Criteria:

* Not placed in an ACS run-or contracted facility enrolled in the study during the study period
* Lack of proficiency in English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-04-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Decreases in Suicidal Ideation Questionnaire (Davis, 1992) and suicide subscale of Massachusetts Youth Screening Instrument (Grisso et al., 2001) | 1 year
  Change in suicide ideation, thoughts, and behaviors
Decreases on Self-Injurious Thoughts and Behaviors Interview (Nock et al., 2007) | 1 year
  Change in self-harm thoughts and behaviors
Decreases on internalizing and externalizing subscales of Massachusetts Youth Screening Instrument (Grisso et al., 2001) | 1 year
  Change in mental health correlates of suicide
Decreased burnout and increased job efficacy on the Professional Quality of Life measure (Stramm, 2016) and the Maslach Burnout Inventory | 1 year
  Change in staff burnout and job efficacy
Change in responses on the Inventory of Depression and Anxiety Symptoms (Watson et al., 2007) | 1 year
  Change in staff mental health
Increased suicide knowledge and response skills from Tennessee's state-wide gatekeeper training (Schut & Lockman, 2013) | 1 year
  Change in suicide knowledge and response skills
Increased self-harm knowledge response skills from Tennessee's state-wide gatekeeper training (Schut & Lockman, 2013) | 1 year
  Change in self-harm knowledge and response skills

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT05658068/ICF_000.pdf